CLINICAL TRIAL: NCT02557178
Title: Home-Based Health Management of COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Seifert (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Mayo Clinic (Other)
Responsible Party: Sponsor-Investigator, Sara Seifert, President, Minnesota HealthSolutions
Organization: Minnesota HealthSolutions (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: R44HL114162-02A1 (NIH); R44HL114162 (NIH)
Record Dates: First submitted 2015-03-03; First posted 2015-09-23 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Activity Monitor plus Health Coaching (Experimental): Device: Actigraph Participants will wear the device daily during weeks 1, 9, and 17. Daily steps and activity will be measured. It will identify if they complete a prescribed exercise regimen. Participants in the intervention condition (wearing the Actigraph) will also receive supportive health coaching to encourage them to exercise.
  Interventions: Behavioral: health coaching
- Control (No Intervention): Device: Actigraph Participants will wear the device daily during weeks 1, 9, and 17. Daily steps and activity will be measured. It will identify if they complete a prescribed exercise regimen.

INTERVENTIONS:
Behavioral: health coaching — Supportive coaching to encourage compliance with prescribed pulmonary rehabilitation.
  Arms: Activity Monitor plus Health Coaching

SUMMARY:
Minnesota HealthSolutions Corporation (MHS) proposes to develop and evaluate a program to motivate and monitor people with chronic obstructive pulmonary disease (COPD) to complete home exercise as part of pulmonary rehabilitation (PR). The proposed system has two components: home-based activity monitoring and health coaching. The investigators will conduct a randomized, wait-list controlled clinical study to evaluate the effects of the activity monitoring system and health coaching on quality of life and daily steps.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of GOLD stage II, III, or IV COPD
* current or previous smoker with at least 10 pack-years of cigarette smoking
* be hospitalized for an exacerbation of COPD

Exclusion Criteria:

* high likelihood of being lost to follow-up or contact
* inability to provide good data or follow commands
* inability to do mild exercise

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-09; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Seifert, MPH, Principal Investigator — Minnesota HealthSolutions
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benzo RP, Ridgeway J, Hoult JP, Novotny P, Thomas BE, Lam NM, V Benzo M, Kramer K, Seifert S. Feasibility of a Health Coaching and Home-Based Rehabilitation Intervention With Remote Monitoring for COPD. Respir Care. 2021 Jun;66(6):960-971. doi: 10.4187/respcare.08580. Epub 2021 Apr 27. PMID 33906954

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 controls off study before completing baseline forms or phone calls (1 withdrew and 1 lost to follow up) 6 intervention participants off study before completing baseline forms or phone calls (5 withdrew and 1 lost to follow up)
Period: Overall Study
Arm/Group | Activity Monitor Plus Health Coaching | Control
Started | 72 | 74
Completed | 56 | 63
Not Completed | 16 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Activity Monitor Plus Health Coaching | Control | Total
Number analyzed (Participants) | 72 | 74 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (8.1) | 68.5 (9.1) | 68.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 75
  Male | 34 | 37 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 70 | 73 | 143
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Physical Activity from ActiGraph [Mean (Standard Deviation); unit: steps] | 3547.3 (1835.8) | 4426.3 (2628.3) | 4016.1 (2326.7)
Quality of Life Physical Summary [Mean (Standard Deviation); unit: units on a scale] — The Chronic Respiratory Disease Questionnaire uses 20 items in four categories to assess quality of life. Physical summary uses the dyspnea and fatigue categories. The items are assessed numerically on a 7-point modified Likert scale. Scores for each category are obtained by adding the scores for the items that make up the category and dividing by the number of items. Physical summary adds the fatigue and dyspnea scores and divides by two; hence, the range for each item, domain, and physical scale is 1 to 7. A minimally important difference is a change in score of 0.5 or more.
  units on a scale | 4.3 (1.2) | 4.2 (1.1) | 4.2 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Daily Steps Between the Intervention and Control Conditions
Description: Number of daily steps as measured by the SenseWear Pro ArmBand, which is an accepted criterion measure for daily physical activity in adults with Chronic Obstructive Pulmonary Disease.
Time Frame: Steps measured at baseline (week 1) and week 9
Population: Data is provided for 119 participants who completed the study.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Activity Monitor Plus Health Coaching | Control
Number analyzed (Participants) | 56 | 63
steps | -344.8 (1657.7) | -975.8 (2596.3)

2. Primary Outcome: Change in Physical Quality of Life Between the Intervention and Control Conditions
Description: Measure Description: The Chronic Respiratory Disease Questionnaire measures physical and emotional aspects with 20 items in four domains/categories. The two domains/categories used for physical summary were dyspnea and fatigue. The items are assessed numerically on a 7-point modified Likert scale (from 1 to 7). Scores are obtained by adding the scores for the items that make up each category and dividing by the number of items. Physical quality of life is obtained by adding the fatigue and dyspnea scores and dividing by two; hence, the score range is from 1 to 7. Higher scores indicate better health-related quality of life. Scores are obtained by adding the scores for the items that make up each category and dividing by the number of items. A minimally important difference is a change in score of 0.5 or more.
Time Frame: Quality of Life measured at baseline (week 1) and week 9
Population: Data is provided for 119 participants who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Activity Monitor Plus Health Coaching | Control
Number analyzed (Participants) | 56 | 63
units on a scale | 0.2 (1.0) | 0.0 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored through the study time frame, an average of 17 weeks per participant.
Arm/Group | Activity Monitor Plus Health Coaching | Control
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/74
Other Adverse Events (participants affected / at risk) | 0/72 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT02557178/Prot_SAP_000.pdf